CLINICAL TRIAL: NCT06197854
Title: Onlay Versus Sublay Hernioplasty in Management of Incisional Hernia
Brief Title: Onlay Versus Sublay Mesh in Incisional Hernia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mark Awny Albeir Saad, Resident doctor, Assiut University
Other Study IDs: Mesh in incisional hernia
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia | interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sublay hernioplasty in incisional hernia: Group that will undergo Sublay hernioplasty in management of incisional hernia
  Interventions: Procedure: Hernioplasty
- Onlay Hernioplasty in incisional hernia: Group that will undergo Onlay hernioplasty in management of incisional hernia
  Interventions: Procedure: Hernioplasty

INTERVENTIONS:
Procedure: Hernioplasty — Surgical hernioplasty

SUMMARY:
Onlay versus Sublay Mesh hernioplasty in management of incisional Hernia Comparative prospective study (Short term outcomes)

DETAILED DESCRIPTION:
Comparison between Short term outcomes (advantages and disadvantages) of sublay and onlay techniques in management of incisional hernia regarding :

* Short term complications (superficial skin infection, seroma formation , recurrence and chronic abdominal discomfort.)
* operative time , hospital stay , difficulty of technique.

ELIGIBILITY:
Inclusion Criteria:

* Surgically Fit patients
* Patients presented with incisional Hernias
* Age between 18 to 60 years
* Cicatrized incisional hernia involving both muscle cutting and muscle splitting incisions

Exclusion Criteria:

* Surgically unfit patients
* Irreducible, obstructed, strangulated hernias
* Other Ventral hernias that not related to surgical incision.
* Huge hernias with wide abdominal wall defect and retracted abdominal wall muscles.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Any patient presenting with incisional hernia for elective hernioplasty that is Surgically Fit and match inclusion critiria
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Short term complications | 1 month
  (Recurrence, Post operative Pain, seroma and skin infection.)

SECONDARY OUTCOMES:
Post operative complications | 1 month
  Superficial skin infection, seroma formation, recurrence and chronic abdominal discomfort.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schlosser KA, Arnold MR, Otero J, Prasad T, Lincourt A, Colavita PD, Kercher KW, Heniford BT, Augenstein VA. Deciding on Optimal Approach for Ventral Hernia Repair: Laparoscopic or Open. J Am Coll Surg. 2019 Jan;228(1):54-65. doi: 10.1016/j.jamcollsurg.2018.09.004. Epub 2018 Oct 22. PMID 30359827
- [Background] Mathes T, Walgenbach M, Siegel R. Suture Versus Mesh Repair in Primary and Incisional Ventral Hernias: A Systematic Review and Meta-Analysis. World J Surg. 2016 Apr;40(4):826-35. doi: 10.1007/s00268-015-3311-2. PMID 26563217
- [Background] Deeken CR, Lake SP. Mechanical properties of the abdominal wall and biomaterials utilized for hernia repair. J Mech Behav Biomed Mater. 2017 Oct;74:411-427. doi: 10.1016/j.jmbbm.2017.05.008. Epub 2017 May 6. PMID 28692907
- [Background] Smietanski M, Bury K, Tomaszewska A, Lubowiecka I, Szymczak C. Biomechanics of the front abdominal wall as a potential factor leading to recurrence with laparoscopic ventral hernia repair. Surg Endosc. 2012 May;26(5):1461-7. doi: 10.1007/s00464-011-2056-8. Epub 2011 Dec 15. PMID 22170318
- [Background] Hawn MT, Gray SH, Snyder CW, Graham LA, Finan KR, Vick CC. Predictors of mesh explantation after incisional hernia repair. Am J Surg. 2011 Jul;202(1):28-33. doi: 10.1016/j.amjsurg.2010.10.011. PMID 21741517
- [Background] Rosen MJ, Bauer JJ, Harmaty M, Carbonell AM, Cobb WS, Matthews B, Goldblatt MI, Selzer DJ, Poulose BK, Hansson BM, Rosman C, Chao JJ, Jacobsen GR. Multicenter, Prospective, Longitudinal Study of the Recurrence, Surgical Site Infection, and Quality of Life After Contaminated Ventral Hernia Repair Using Biosynthetic Absorbable Mesh: The COBRA Study. Ann Surg. 2017 Jan;265(1):205-211. doi: 10.1097/SLA.0000000000001601. PMID 28009747
- [Background] Cobb WS, Warren JA, Ewing JA, Burnikel A, Merchant M, Carbonell AM. Open retromuscular mesh repair of complex incisional hernia: predictors of wound events and recurrence. J Am Coll Surg. 2015 Apr;220(4):606-13. doi: 10.1016/j.jamcollsurg.2014.12.055. Epub 2015 Jan 28. PMID 25797746